CLINICAL TRIAL: NCT01415063
Title: Radiofrequency Ablation Combined With Transcatheter Arterial Chemoembolization Versus Radiofrequency Ablation Alone for Recurrent Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Cancer Center, Sun Yat-sen University, Cancer Center, Sun Yat-sen University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HCC-0013
Record Dates: First submitted 2011-08-10; First posted 2011-08-11 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-02

CONDITIONS: Hepatocellular Carcinoma; RFA; TACE
Keywords: Hepatocellular Carcinoma; RFA; TACE
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RFA (Experimental): For RFA, we used a commercially available system with a 375-KHz computer-assisted radiofrequency generator (Elektrotom HiTT 106, Berchtold, Medizinelektronik, Germany) and an open-perfused electrode (Berchtold, Tuttlingen, Germany) of 15 cm (or 20 cm), 14 Ga, and a 15 mm (or 20 mm) active electrode tip with microbores.
  Interventions: Procedure: TACE-RFA
- TACE-RFA (Experimental): TACE first, then RFA within 2 weeks
  Interventions: Procedure: RFA

INTERVENTIONS:
Procedure: RFA — For RFA, we used a commercially available system with a 375-KHz computer-assisted radiofrequency generator (Elektrotom HiTT 106, Berchtold, Medizinelektronik, Germany) and an open-perfused electrode (Berchtold, Tuttlingen, Germany) of 15 cm (or 20 cm), 14 Ga, and a 15 mm (or 20 mm) active electrode tip with microbores.
  Arms: TACE-RFA
Procedure: TACE-RFA — TACE first, then RFA within 2 weeks
  Arms: RFA

SUMMARY:
The combination of transcatheter arterial chemoembolization (TACE) with RFA has also reported to be an effective treatment for HCC. Studies have shown TACE combined RFA to have better efficacy than RFA for medium-sized HCC (3-5 cm) and multiple-tumor HCC, but not for small HCC (≤3 cm). However, to our knowledge, there have not been any prospective studies to assess whether TACE combined sequentially with RFA is more effective than RFA alone for the treatment of HCC recurrence after curative treatment. We hypothesized that the combination of TACE and RFA might result in better patient survival than RFA alone. Thus, the purpose of this study was to prospectively compare the effects of sequential TACE-RFA with RFA alone for the treatment of recurrent HCC. Recurrent HCC in this study was defined as new tumors in the remnant liver, distant from the resection or ablation site after curative treatment of RFA or hepatectomy.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the fifth most common cancer in the world. Partial hepatectomy and liver transplantation are considered to be standard curative therapies for HCC. When surgery is not possible, percutaneous ablation is usually considered to be alternative treatments for HCC . Recurrence is the most frequent serious adverse event observed during the follow-up of HCC patients treated for cure. Repeat hepatectomy is an effective treatment for HCC recurrence, with a 5-year survival rate of 19.4 to 56%. Unfortunately, repeat hepatectomy can be performed only in a small proportion of patients with HCC recurrence (10.4 to 31%), either because of the poor functional liver reserve or because of widespread recurrence.(15, 17, 18) Radiofrequency ablation (RFA) has been considered to be one of the most effective percutaneous ablations for early-stage HCC in patients with or without surgical prospects . Studies using RFA to treat HCC recurrence after hepatectomy have reported a 3-year survival rate of 62% to 68%, which is comparable to those achieved by surgery. RFA is particularly suitable to treat HCC recurrence after hepatectomy because these tumors are usually detected when they are small, and because RFA causes the least deterioration of liver function in the patients. RFA is also effective for managing HCC recurrence after initial treatment of RFA. Clinical data have shown that, after repeated RFA, the estimated 3-and 5-year overall, and disease-free survival rates for patients with HCC recurrence were 67.0% and 40.1% and 68.0 and 38.0%, respectively.Therefore, we considered RFA to be an effective treatment for HCC recurrence after curative treatment.

The combination of transcatheter arterial chemoembolization (TACE) with RFA has also reported to be an effective treatment for HCC. Studies have shown TACE combined RFA to have better efficacy than RFA for medium-sized HCC (3-5 cm) and multiple-tumor HCC, but not for small HCC (≤3 cm). However, to our knowledge, there have not been any prospective studies to assess whether TACE combined sequentially with RFA is more effective than RFA alone for the treatment of HCC recurrence after curative treatment. We hypothesized that the combination of TACE and RFA might result in better patient survival than RFA alone. Thus, the purpose of this study was to prospectively compare the effects of sequential TACE-RFA with RFA alone for the treatment of recurrent HCC. Recurrent HCC in this study was defined as new tumors in the remnant liver, distant from the resection or ablation site after curative treatment of RFA or hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 - 75 years;
2. Distant recurrence of HCC after initial curative treatment (including initial RFA or hepatectomy);
3. no other treatment received except for the initial RFA or hepatectomy;
4. Single tumor less than 4cm in diameter;
5. lesions visible on ultrasound and with an acceptable and safe path between the lesion and the skin as shown on ultrasound;
6. no severe coagulation disorders (prothrombin activity < 40% or a platelet count of < 40,000 / mm3;
7. Eastern Co-operative Oncology Group performance(ECOG) status 0 -

Exclusion Criteria:

1. the presence of vascular invasion or extrahepatic spread on imaging;
2. a Child-Pugh class C liver cirrhosis or evidence of hepatic decompensation including ascites, severe coagulation disorders (prothrombin activity < 40% or a platelet count of < 40,000 / mm3), esophageal or gastric variceal bleeding or hepatic encephalopathy;
3. an American Society of Anesthesiologists (ASA) score ≥ 3

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-02; Primary Completion 2013-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
overall survival | 1 year

SECONDARY OUTCOMES:
disease-free survival | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center, Sun Yat-set University, Guangzhou, Guangdong, China